CLINICAL TRIAL: NCT04477941
Title: The Association Between Parents' Stress and Feeding Styles and Practices: Systematic Review and Meta-analysis of Observational Studies
Brief Title: Systematic Review of Parents' Stress and Feeding Styles and Practices
Status: Completed | Type: Observational
Sponsor: Mathilda Vandenheuvel (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Mathilda Vandenheuvel, Staff physician, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 1000058039
Record Dates: First submitted 2020-07-04; First posted 2020-07-20 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Parent-Child Relations; Stress; Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parents' mental health contributes to their feeding practices how they perceive and respond to their children's behavior. Suboptimal feeding practices may promote dysfunctional eating behaviours in children and contribute to children's weigh. The purpose of this review is to identify existing literature on the association between parents' stress and their feeding styles and practices

DETAILED DESCRIPTION:
Background:

Feeding is a central aspect of parenting that involves interactions between parents and their children. Those feeding interaction influence children's eating behaviors during a sensitive period of growth and cognitive development. Parents' feeding styles and parents' feeding practices are terms that have been used to describe feeding interactions between parents and their children. Previous research have found that parents' feeding styles and feeding practices are associated with different children's outcomes (e.g. growth, weight).Throughout literature, the terms of parents' feeding styles and feeding practices have been used interchangeably.

Parenting styles can be defined as attitudes or an emotional climate that characterizes the parents' approach and interaction with their children across different domains of parenting. Those domains can be characterized based on demandingness (defined as behavioral control over the child) and responsiveness (defined as warmth and supportiveness for the child). Based on those domains there are four parenting styles: authoritative, authoritarian, indulgent and neglectful. An authoritative parenting style can be characterized as a style associated with a high level of responsiveness and demandingness to the child. As for the authoritarian parenting style can be defined as style with low responsiveness and high demandingness. Whereas the indulgent parenting style can be characterized as a style with high responsiveness and engagement with the child but with low demandingness. Finally, an uninvolved parenting style is defined as a style with both low responsiveness and low demandingness.

Parenting feeding styles can be defined as attitudes or an emotional climate that characterizes the parents' approach with their children during feeding interaction. Feeding styles are a sub-category of parenting styles with similar domains of responsiveness and demandingness applied within a feeding context. For instance, an authoritarian feeding style is where a parent supports and encourages their child eating with directives and rules regardless to the child's preferences, whereas a parent with an authoritative feeding style a parent encourages eating with a non-directive approach and is responsive to the child's preferences and needs.

Parents' feeding practices concept refers to the strategies and techniques parents may employ to maintain or control the feeding context such as when, what or how much their children eat. Feeding practices are intended specific behaviors parents use to influence their children's eating and differ based on parents' perceptions and beliefs of how to achieve optimal growth for their children. For instance, a parent could limit access to certain food types to control his/her child's weight, or force feed the child to increase his/her weight. Different feeding practices have been discussed in literature such as restriction of certain food types, pressuring to eat, or using food as a reward. Feeding practices have been associated with weight and eating behaviors in children. Ventura and Birch argue that parental feeding practices are a response to a child's behaviour rather than a parental trait.Moreover, parental feeding style can be consistent, or found within a parent, but parental feeding practices can be different depending on different factors such as a child's weight and temperament.

Parents' mental health influence parents' feeding style and practices.The World Health Organization (WHO) defines mental health as "a state of well-being in which individual realizes his or her own abilities, can cope with the normal stresses of life, can work productively and fruitfully, and is able to make a contribution to his or her community". Caregivers' mental health problems are considered to be a major public health challenge worldwide. Parents' mental health, such as stress and depression, influences how they perceive their children's behavior, as well as how they interpret and respond to their child behaviors. In a study by Hurley et al, they found that mothers who experienced more symptoms of stress, depression and anxiety were more likely to engage in non-responsive feeding practices. In another study by Swyden et al, they found an association between mothers with a high level of stress and restrictive feeding practices such as restricting the amount and type of food been consumed.

Stress in general can be characterized as the ability to cope with challenges, or an emotional or behavioral response an individual may experience toward an unpleasant event. While parenting stress can be conceptualized as psychological distress experienced by parents as a response to their efforts to meet parenting demands. Different studies have examined parents' stress (either general stress or parenting stress) in association with feeding style and practices of parents, child weight and eating behaviours. For instant, in a cross-sectional study, mothers who reported a high level of stress symptoms were more likely to engage in forceful, controlling and restriction feeding practices. In another cross-sectional study by Hughes et al, the relationship between parental emotional distress and feeding style in low-income parents with preschool children was examined. They reported that parents with uninvolved feeding style had a high level of parenting stress compared to parents with other feeding styles: authoritative- authoritarian and indulgent. These results support the claim that there is a relationship between parents' stress and their feeding styles and/or practices.

Objective:

The primary objective of this systematic review and met-analysis is to summarize existing literature on the association between parents' stress (both parenting and general stress) and parents' feeding styles and practices (both parents' emotional climate and strategies applied in the context of feeding).

Design:

This systematic review and meta-analysis will be conducted according to the Cochran Handbook for Systematic Reviews of Interventions and the results will be reported according to Meta-Analysis of Observational Studies in Epidemiology (MOOSE) guidelines and Preferred Reporting Items of Systematic Reviews and Meta-Analyses (PRISMA) guidelines.

Data Sources:

The investigators will search the following databases: MEDLINE, EMBASE, and PSYCHINFO (accessed via Ovid), CINAHL (accessed via Ebsco). The authors will apply appropriate search strategy through database. Searches will be supplemented with manual searches of references of included publications.

Data Extraction:

Two or more investigators will independently extract relevant data and assess risk of bias. First, title and abstract of identified studies will be screened for eligibility. Second, full texts will be examined in detail based on eligibility criteria outlined above. Third, references of all considered articles will be screened for any potentially eligible studies that were not captured in the search strategy. Any disagreement between the reviewers will be resolved by author (MV). For missing data, authors of primary publication will be contacted. Risk of bias for observational studies will be assessed using the Newcastle Ottawa Scale. As for cross-sectional studies, risk of bias will be assessed using the National Institutes of Health "Quality assessment tool for observational cohort and cross-sectional studies".

Data synthesis and statistical analysis:

The extracted data from included studies (e.g., participants' characteristics, exposure, outcomes, results and direction of association) will be used to build an evidence table. Also, if sufficient studies are identified and variability is low, data from included studies will be pooled using the generic inverse variance method. A random-effect model will be used to determine the association between parents' stress and their feeding styles.This will be done under the assumption that the true effects are normally distributed. Fixed-effects models will be used only where there are <5 included associations.

Assessment of heterogeneity:

The investigators will evaluate heterogeneity by estimating the variance between studies using Cochran Q statistic and quantified by the I2 statistic. The Cochran's Q test is obtained by the weighted sum of the squared differences of the observed effect in each study minus the fixed summary effect. The I2 statistic describes the percentage of variability in the effect estimate that is not due to chance and (I2 >= 50%) indicates a substantial heterogeneity with a p-value of <0.1 as a statistically significant level. To explore sources of heterogeneity, investigators will conduct sensitivity analyses in which each study is systematically removed. If >=10 studies are available, potential sources of heterogeneity by a priori subgroup analyses will be explored. The investigators will conduct subgroup analyses that will depend on identified studies; determined by study design (prospective or retrospective), follow-up time, setting (developed or developing countries), socio-demographic characteristics, sample size and adjustment for confounding variables (i.e., gender, education and history of mental health). If >=10 studies are available, publication bias will be assessed by an inspection of funnel plots and tested using the Egger and Begg test. If publication bias is suspected, the Duval and Tweedie trim and fill method will be applied to adjust for funnel plot asymmetry by imputing missing study data.

Evidence Assessment:

Two reviewers will independently assess the quality and strength of included studies using the Grading of Recommendation Assessment, Development and Evaluation (GRADE) system.

Observation studies start at low-quality evidence and can be downgraded or upgraded based on the following criteria:

1. Criteria to downgrade evidence: risk of bias, inconsistency, indirectness, imprecision and publication bias.
2. Criteria to upgrade evidence: large effect size, attenuation by all plausible confounding effects and dose-response gradient.

Differences will be reconciled by consensus.

ELIGIBILITY:
Inclusion Criteria:

* Measurement of Feeding styles and/ or practices measurement (self - report assessment and / or observational assessment)
* Measurement of parent's stress (using assessment tools for stress in the study)
* Observational design, (prospective and retrospective) with no follow-up time restrictions
* Cross-sectional design
* Breastfeeding and complementary feeding studies

Exclusion Criteria:

* Animal studies
* Review studies
* Post-partum depression

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of children (birth- 5 years)
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
the correlation between parents' stress and their feeding styles and practices | follow up, up to 20 years
  The difference in feeding style and practices in different levels of parents' stress expressed in mean difference or standardized mean difference (if different assessment tools were used in included studies)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Nordang S, Shoo T, Holmboe-Ottesen G, Kinabo J, Wandel M. Women's work in farming, child feeding practices and nutritional status among under-five children in rural Rukwa, Tanzania. Br J Nutr. 2015 Nov 28;114(10):1594-603. doi: 10.1017/S0007114515003116. Epub 2015 Oct 5. PMID 26435007
- [Background] Shloim N, Edelson LR, Martin N, Hetherington MM. Parenting Styles, Feeding Styles, Feeding Practices, and Weight Status in 4-12 Year-Old Children: A Systematic Review of the Literature. Front Psychol. 2015 Dec 14;6:1849. doi: 10.3389/fpsyg.2015.01849. eCollection 2015. PMID 26696920
- [Background] Blissett J. Relationships between parenting style, feeding style and feeding practices and fruit and vegetable consumption in early childhood. Appetite. 2011 Dec;57(3):826-31. doi: 10.1016/j.appet.2011.05.318. Epub 2011 May 27. PMID 21651932
- [Background] Ventura AK, Birch LL. Does parenting affect children's eating and weight status? Int J Behav Nutr Phys Act. 2008 Mar 17;5:15. doi: 10.1186/1479-5868-5-15. PMID 18346282
- [Background] Faith MS, Scanlon KS, Birch LL, Francis LA, Sherry B. Parent-child feeding strategies and their relationships to child eating and weight status. Obes Res. 2004 Nov;12(11):1711-22. doi: 10.1038/oby.2004.212. PMID 15601964
- [Background] Thompson AL, Adair LS, Bentley ME. Pressuring and restrictive feeding styles influence infant feeding and size among a low-income African-American sample. Obesity (Silver Spring). 2013 Mar;21(3):562-71. doi: 10.1002/oby.20091. PMID 23592664
- [Background] p6rwood RL, Schoelmerich A, Schulze PA, Gonzalez Z. Cultural differences in maternal beliefs and behaviors: a study of middle-class Anglo and Puerto Rican mother-infant pairs in four everyday situations. Child Dev. 1999 Jul-Aug;70(4):1005-16. doi: 10.1111/1467-8624.00073. PMID 10446732
- [Background] Galderisi S, Heinz A, Kastrup M, Beezhold J, Sartorius N. Toward a new definition of mental health. World Psychiatry. 2015 Jun;14(2):231-3. doi: 10.1002/wps.20231. No abstract available. PMID 26043341
- [Background] Hurley KM, Black MM, Papas MA, Caulfield LE. Maternal symptoms of stress, depression, and anxiety are related to nonresponsive feeding styles in a statewide sample of WIC participants. J Nutr. 2008 Apr;138(4):799-805. doi: 10.1093/jn/138.4.799. PMID 18356338
- [Background] Swyden K, Sisson SB, Morris AS, Lora K, Weedn AE, Copeland KA, DeGrace B. Association Between Maternal Stress, Work Status, Concern About Child Weight, and Restrictive Feeding Practices in Preschool Children. Matern Child Health J. 2017 Jun;21(6):1349-1357. doi: 10.1007/s10995-016-2239-y. PMID 28138826
- [Background] Hackie M, Bowles CL. Maternal perception of their overweight children. Public Health Nurs. 2007 Nov-Dec;24(6):538-46. doi: 10.1111/j.1525-1446.2007.00666.x. PMID 17973731
- [Background] Barroso NE, Hungerford GM, Garcia D, Graziano PA, Bagner DM. Psychometric properties of the Parenting Stress Index-Short Form (PSI-SF) in a high-risk sample of mothers and their infants. Psychol Assess. 2016 Oct;28(10):1331-1335. doi: 10.1037/pas0000257. Epub 2015 Nov 23. PMID 26595220
- [Background] Bornstein MH. Handbook of parenting. 2nd ed. Mahwah, N.J.: Erlbaum; 2002.
- [Background] Baker-Henningham H, Hamadani JD, Huda SN, Grantham-McGregor SM. Undernourished children have different temperaments than better-nourished children in rural Bangladesh. J Nutr. 2009 Sep;139(9):1765-71. doi: 10.3945/jn.109.106294. Epub 2009 Jul 15. PMID 19605526
- [Background] Hughes SO, Power TG, Liu Y, Sharp C, Nicklas TA. Parent emotional distress and feeding styles in low-income families. The role of parent depression and parenting stress. Appetite. 2015 Sep;92:337-42. doi: 10.1016/j.appet.2015.06.002. Epub 2015 Jun 4. PMID 26050915
- [Background] Cumpston M, Li T, Page MJ, Chandler J, Welch VA, Higgins JP, Thomas J. Updated guidance for trusted systematic reviews: a new edition of the Cochrane Handbook for Systematic Reviews of Interventions. Cochrane Database Syst Rev. 2019 Oct 3;10(10):ED000142. doi: 10.1002/14651858.ED000142. No abstract available. PMID 31643080
- [Background] Stroup DF, Berlin JA, Morton SC, Olkin I, Williamson GD, Rennie D, Moher D, Becker BJ, Sipe TA, Thacker SB. Meta-analysis of observational studies in epidemiology: a proposal for reporting. Meta-analysis Of Observational Studies in Epidemiology (MOOSE) group. JAMA. 2000 Apr 19;283(15):2008-12. doi: 10.1001/jama.283.15.2008. PMID 10789670
- [Background] Shamseer L, Moher D, Clarke M, Ghersi D, Liberati A, Petticrew M, Shekelle P, Stewart LA; PRISMA-P Group. Preferred reporting items for systematic review and meta-analysis protocols (PRISMA-P) 2015: elaboration and explanation. BMJ. 2015 Jan 2;350:g7647. doi: 10.1136/bmj.g7647. PMID 25555855
- [Background] DerSimonian R, Laird N. Meta-analysis in clinical trials. Control Clin Trials. 1986 Sep;7(3):177-88. doi: 10.1016/0197-2456(86)90046-2. PMID 3802833
- [Background] Cochran WG. The Combination of Estimates from Different Experiments. Biometrics. 1954;10:101-29.
- [Background] Higgins JP, Thompson SG, Deeks JJ, Altman DG. Measuring inconsistency in meta-analyses. BMJ. 2003 Sep 6;327(7414):557-60. doi: 10.1136/bmj.327.7414.557. PMID 12958120
- [Background] Egger M, Davey Smith G, Schneider M, Minder C. Bias in meta-analysis detected by a simple, graphical test. BMJ. 1997 Sep 13;315(7109):629-34. doi: 10.1136/bmj.315.7109.629. PMID 9310563
- [Background] Begg CB, Mazumdar M. Operating characteristics of a rank correlation test for publication bias. Biometrics. 1994 Dec;50(4):1088-101. PMID 7786990
- [Background] Shi L, Lin L. The trim-and-fill method for publication bias: practical guidelines and recommendations based on a large database of meta-analyses. Medicine (Baltimore). 2019 Jun;98(23):e15987. doi: 10.1097/MD.0000000000015987. PMID 31169736
- [Background] Guyatt GH, Oxman AD, Vist GE, Kunz R, Falck-Ytter Y, Alonso-Coello P, Schunemann HJ; GRADE Working Group. GRADE: an emerging consensus on rating quality of evidence and strength of recommendations. BMJ. 2008 Apr 26;336(7650):924-6. doi: 10.1136/bmj.39489.470347.AD. PMID 18436948
- [Background] Bennett IM, Schott W, Krutikova S, Behrman JR. Maternal mental health, and child growth and development, in four low-income and middle-income countries. J Epidemiol Community Health. 2016 Feb;70(2):168-73. doi: 10.1136/jech-2014-205311. Epub 2015 Sep 10. PMID 26359503